CLINICAL TRIAL: NCT06684197
Title: The Impact of a Dexmedetomidine Perfusion on Intraoperative Remifentanil Consumption: a Randomized Controlled Trial
Brief Title: The Impact of a Dexmedetomidine Perfusion on Intraoperative Remifentanil Consumption
Acronym: DEXREM
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ciusss de L'Est de l'Île de Montréal (Other)
Responsible Party: Principal Investigator, Olivier Verdonck, MD, MSc, Clinical Assistant Professor, Head of Department of Anesthesiology and Pain Medecine, Maisonneuve-Rosemont Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CAR 2025-3856
Record Dates: First submitted 2024-11-08; First posted 2024-11-12 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-11

CONDITIONS: Dexmedetomidine; Total Intravenous Anesthesia; Remifentanil Consumption; Remifentanil; Laparoscopic Abdominal Surgery
MeSH Terms: interventions — Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dexmedetomidine (Active Comparator): Dexmedetomidine 0.5 mcg/kg (adjusted body weight) ; Administered via infusion pump (Smith Medical Medfusion® 4000 Syringe Infusion Pump) delivered over 10 minutes during induction of general anesthesia, followed by dexmedetomidine 0.5 mcg.kg-1.h-1 (maximum dose: 2.5mcg.kg-1)
  Interventions: Drug: Dexmedetomidine
- Placebo - Normal Saline (Placebo Comparator): Normal saline in volume equivalent of dexmedetomidine dose according to patient weight ; Administered via infusion pump (Smith Medical Medfusion® 4000 Syringe Infusion Pump) so that the full dose is delivered is equivalent to a maximum dose of 2.5mcg.kg-1 of dexemedetomidine
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dexmedetomidine — Intravenous dexmedetomidine will be given as a bolus (0.5 μg.kg-1) over 10 minutes. A perfusion of 0.5 mcg.kg-1.h-1 of dexmedetomidine will be programmed and maintained up until the pneumoperitoneum is deflated or up until a total dose of 2.5μg.kg-1 has been administered.
  Arms: Dexmedetomidine
Drug: Placebo — Saline will be used instead of dexmedetomidine
  Arms: Placebo - Normal Saline

SUMMARY:
Opioids analgesic are the gold standard for intraoperative pain management. Their short- and long-term adverse effect motivate anesthesiologists to explore opioid sparing strategies. Dexmedetomidine is a highly selective α2 adrenergic receptor agonist that could help minimize opioid consumption both intraoperative and postoperative due to its sedative, analgesic and sympatholytic properties. This new randomized controlled trial (RCT) will answer the question whether an intraoperative dexmedetomidine infusion compared to placebo has a clinically significant impact on intraoperative remifentanil consumption during a laparoscopic abdominal elective surgery.

DETAILED DESCRIPTION:
Opioids analgesic have been used for intraoperative pain management for decades. They are the gold standard for pain relief due to their high efficacy. However, the short- and long-term adverse effects of opioids motivate anesthesia teams to explore opioid sparing strategies employing a combination of analgesics and adjuvants via continuous infusions. Opioid tolerance and opioid-induced hyperalgesia can lead to dose escalation of prescribed opioids and poor pain control.

Dexmedetomidine is a highly selective α2 adrenergic receptor agonist that could help minimize opioid consumption both intraoperative and postoperative due to its sedative, analgesic and sympatholytic properties. Other post-procedure applications such as reduction of cough, agitation and shivering have been described.

Many trials have studied the impact of intraoperative dexmedetomidine on post-operative pain scores, post-operative opioids consumption and common side effects compared with a remifentanil intraoperative infusion. One randomized controlled trial studied the impact of a 30 min dexmedetomidine infusion on intraoperative remifentanil consumption in ASA 1-2 patients undergoing maxillofacial or cervicofacial surgeries. They found a clinically meaningful reduction of 33% of remifentanil consumption at 120 minutes in the dexmedetomidine group. This trial aims to demonstrate a similar reduction when extending to ASA 3 patients undergoing laparoscopic surgery. Furthermore, the investigators aim to evaluate patients' recovery and pain status 24h after the surgery which hasn't been done before in the context of joint dexmedetomidine and remifentanil infusion. The investigators hypothesize that patients of the dexmedetomidine infusion group will require less intraoperative remifentanil to keep the NOL-index into the prespecified range. In the PACU, lower pain score et less opioids requirements are anticipated.

ELIGIBILITY:
Inclusion Criteria:

* ASA 1-3
* Laparascopic surgery (including general surgery, gynecology, urology) a small abdominal incision (less than 5 cm) will be tolerated.

Exclusion Criteria:

* Patient refusal
* Chronic use of opioids
* Allergy to medication used in the trial
* Pregnant or breastfeeding women
* Contraindications to dexmedetomidine (Bradycardia, arrythmia or pace- maker, severe ventricular dysfunction)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2024-11 (Estimated); Primary Completion 2025-11 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Remifentanil consumption expressed in mcg.kg-1.h-1 | From induction of anesthesia to end of surgery
  Compare remifentanil consumption when using an intraoperative dexmedetomidine infusion (bolus of 0.5mcg.kg-1, than infusion of 0.5 mcg.kg-1.h-1, with a maximum dose of 2.5 mcg.kg-1) versus placebo (normal saline)

SECONDARY OUTCOMES:
Total intraoperative propofol consumption (mg.kg-1.h-1) | From induction of anesthesia to end of surgery
  Compare the total intraoperative propofol consumption during anesthesia, to maintien BIS values between 40-60
Mean intraoperative blood pressure | From induction of anesthesia to end of surgery
  Compare intraoperative blood pressure in both groups (mmHg)
Number of intraoperative episodes of high/low blood pressure | From induction of anesthesia to end of surgery
  Compare episodes of high blood pressure (defined as + 20% of patient's baseline) ans episodes of low blood pressure (defined as - 20% of patient's baseline) between both groups
Number of episodes of intraoperative tachy-/bradycardia | From induction of anesthesia to end of surgery
  Compare episodes of tachycardia (defined as > 100 bpm) and episodes of bradycardia (defined as < 45 bpm) between both groups
Total intraoperative dose of vasopressors | From induction of anesthesia to end of surgery
  Compare the intraoperative requirements of norepinephrine, ephedrine, glycopyrrolate and atropine.
intraoperative NOL index | From intubation to end of surgery
  compare the percentage of time during the intraoperative period for which the NOL index will be above the pain threshold of 25
Time for extubation (in minutes) | From end of surgery to extubation
  Compare the time for extubation
Morphine equivalent consumption in the post anesthesia care unit (PACU) | From PACU admission to discharge from PACU (Aldrete Score >=9 / 10)
  Compare total amount of morphine equivalent given in the post anesthesia care unit (mesured in mg)
Pain scores using visual analogue scale (VAS) in PACU | From PACU admission to discharge from PACU (Aldrete Score >=9 / 10)
  Compare pain scores using VAS in PACU
Adverse events in PACU | From PACU admission to discharge from PACU (Aldrete Score >=9 / 10)
  Compare adverse events in PACU: hypotension, bradycardia and post-operative nausea and vomiting (PONV)
Lenght of stay in PACU (in minutes) | From PACU admission to discharge
  Compare total time for readiness for discharge from PACU between groups assessed by recovery scores (Aldrete's modified score and Maisonneuve-Rosemont PACU score)
Pain scores using numeric rating scale (NRS) 24h post-op | post-op day 1
  Compare pain score between both groups 24h post-op
Quality of recovery (QoR) index 24h post-op | post-op day 1
  Compare Quality of recovery (QoR) index 24h post-op
Mean intraoperative heart rate | From induction of anesthesia to end of surgery
  Compare intraoperative heart rate in both groups (beats per minute)

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Maisonneuve-Rosemont, Montreal, Quebec, Canada

REFERENCES:
- [Result] Coeckelenbergh S, Doria S, Patricio D, Perrin L, Engelman E, Rodriguez A, Di Marco L, Van Obbergh L, Estebe JP, Barvais L, Kapessidou P. Effect of dexmedetomidine on Nociception Level Index-guided remifentanil antinociception: A randomised controlled trial. Eur J Anaesthesiol. 2021 May 1;38(5):524-533. doi: 10.1097/EJA.0000000000001402. PMID 33259449